CLINICAL TRIAL: NCT01824901
Title: A Phase I/Randomized Phase II Study of Docetaxel With or Without AZD4547 in Recurrent FGFR1-Amplified Squamous Non-Small Cell Lung Cancer
Brief Title: Docetaxel With or Without FGFR Inhibitor AZD4547 in Treating Patients With Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2512; NCI-2012-01940 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA021115 (NIH); E2512 (Other: ECOG-ACRIN Cancer Research Group)
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Squamous Cell Lung Cancer
Keywords: AZD4547; recurrent non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; AZD4547

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase I (Experimental): Patients receive docetaxel IV over 60 minutes on day 1 and FGFR inhibitor AZD4547 PO BID on days 2-15 of course 1 and days 1-14 of all subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: AZD4547
- Arm I (docetaxel; phase II step I) (Experimental): Patients receive docetaxel IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who experience progressive disease may then register to step II treatment and receive FGFR inhibitor AZD4547 PO BID on days 1-14.
  Interventions: Drug: docetaxel
- Arm II (docetaxel and AZD4547; phase II step I) (Experimental): Patients receive docetaxel IV over 60 minutes on day 1 and FGFR inhibitor AZD4547 PO BID on days 1-14. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: AZD4547
- Phase II step II (Experimental): Patients receive FGFR inhibitor AZD4547 PO BID on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: AZD4547

INTERVENTIONS:
Drug: docetaxel — Given IV
  Other Names: Taxotere; NSC 628503
  Arms: Arm I (docetaxel; phase II step I); Arm II (docetaxel and AZD4547; phase II step I); Phase I
Drug: AZD4547 — Given PO
  Other Names: NSC 765338
  Arms: Arm II (docetaxel and AZD4547; phase II step I); Phase I; Phase II step II

SUMMARY:
This randomized phase I/II trial studies the side effects and best dose of fibroblast growth factor receptor (FGFR) inhibitor AZD4547 when given with docetaxel and to see how well it works in treating patients with recurrent non-small cell lung cancer. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. FGFR inhibitor AZD4547 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether docetaxel and FGFR inhibitor AZD4547 are more effective when given together or separately.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determination of a recommended phase II dose for the combination of docetaxel and AZD4547 (FGFR inhibitor AZD4547). (Phase I) II. Estimation and comparison of progression-free survival (PFS) of each treatment arm. (Phase II)

SECONDARY OBJECTIVES:

I. Pharmacokinetic evaluation of docetaxel with or without concomitant AZD4547. Pharmacokinetic evaluation of AZD4547 with concomitant docetaxel. (Phase I) II. Safety assessment and toxicity characterization of the combination. (Phase I) III. Initial assessment of clinical activity of the combination. (Phase I) IV. Response rate. (Phase II) V. Overall survival. (Phase II) VI. Estimation of response to single agent AZD4547 among patients who crossover from single agent docetaxel. (Phase II) VII. Further safety assessment and toxicity characterization of AZD4547 alone and in combination with docetaxel. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of FGFR inhibitor AZD4547 followed by a randomized phase II study.

PHASE I:

Patients receive docetaxel intravenously (IV) over 60 minutes on day 1 and FGFR inhibitor AZD4547 orally (PO) twice daily (BID) on days 2-15 of course 1 and days 1-14 of all subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PHASE II, STEP I: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive docetaxel IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who experience progressive disease may then receive FGFR inhibitor AZD4547 PO BID on days 1-14.

ARM II: Patients receive docetaxel IV as in Arm I and FGFR inhibitor AZD4547 PO BID on days 1-14.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PHASE II, STEP II:

Patients receive FGFR inhibitor AZD4547 PO BID on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 years.

This study opened to accrual on September 19, 2013 and was suspended to accrual on January 29, 2014 after each of the first two patients had been registered to the first dose level of the phase I and experienced dose limiting toxicities (DLTs) during week 1 of cycle 1. The study was subsequently terminated on April 17, 2014 after having met the predefined criteria for closure per the phase I study design.

ELIGIBILITY:
Phase I:

Inclusion Criteria:

* All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
* Women of childbearing potential and sexually active males must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Measurable or non-measureable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; baseline measurements and evaluations of all sites of disease must be obtained =< 4 weeks prior to registration
* Histologically or pathologically confirmed squamous NSCLC; patients whose tumors contain mixed NSCLC histologies are eligible if squamous morphology is predominant; mixed tumors with small cell anaplastic elements are not eligible
* Life expectancy >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
* Adequate organ and marrow function
* Mean resting corrected QT interval (QTc) < 470 msec obtained from 3 consecutive electrocardiograms

Exclusion Criteria:

* Pregnant or breast-feeding women
* Clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiogram (ECG) e.g. complete left bundle branch block, third degree heart block
* Factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
* Prior treatment with docetaxel (except in the adjuvant setting), or AZD4547
* Prior treatment with any other chemotherapy, immunotherapy or anticancer agents within 2 weeks prior to registration
* Current evidence or previous history of retinal pigmented epithelium detachment (RPED)
* Previous laser treatment or intra-ocular injection for treatment of macular degeneration
* Current evidence or previous history of dry or wet age-related macular degeneration
* Current evidence or previous history of retinal vein occlusion (RVO)
* Current evidence or previous history of retinal degenerative diseases (e.g. hereditary)
* Current evidence or previous history of any other clinically relevant chorioretinal defect
* Uncontrolled brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD4547, docetaxel or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the investigational drug, previous significant bowel resection, or any other significant gastrointestinal disorder that could, in the opinion of the Investigator, interfere with the absorption of AZD4547
* Major surgical procedure within 3 weeks prior to registration
* Grade 3 or higher peripheral neuropathy, as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE),version 4.02
* Known hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Known human immunodeficiency virus (HIV) with cluster of differentiation (CD)4 count is =< 200 cell/mm^3 or receiving antiretroviral therapy due to potential unfavorable interactions of the agents with the study treatment
* Receiving any other investigational agents while on study
* Medications that are potent inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4), cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8), cytochrome P450, family 2, subfamily D, polypeptide 6 (CYP2D6), or substrates of CYP3A4 prior to the first dose of study treatment

Phase II pre-registration:

* Patient must have paraffin-embedded tumor specimen available for submission for determination of fibroblast growth factor receptor 1(FGFR1) amplification status

Phase II Step I - Randomization:

* Besides the eligibility criteria in Step I, patient must have positive tumor FGFR1 gene amplification (score FISH6) as determined by an AstraZeneca approved central laboratory.

Phase II Step II:

Inclusion Criteria:

* Patient was randomized to docetaxel only on step 1 and progressed per RECIST v1.1 criteria; registration to step 2 must occur within 4 weeks of confirmation/determination of disease progression
* Confirmed measurable disease based on RECIST 1.1; baseline measurements and evaluations of all sites of disease must be obtained =< 4 weeks prior to registration

Exclusion Criteria:

* Pregnant or breast-feeding women

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-01-15 (Actual); Primary Completion 2014-07-09 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rudin, Principal Investigator — Eastern Cooperative Oncology Group
Locations (5):
- United States (5):
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Eastern Cooperative Oncology Group (ECOG) Research Base, Brookline, Massachusetts
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened to accrual on September 19, 2013, accrued its first patient on January 15, 2014, and was suspended to accrual on January 29, 2014 after each of the first two patients had been registered to the first dose level of the phase I and experienced DLTs. The study was subsequently closed on April 17, 2014 after having met the predefined criteria for closure per study design.
Period: Overall Study
Arm/Group | Phase I | Arm I (Docetaxel; Phase II Step I) | Arm II (Docetaxel and AZD4547; Phase II Step I) | Phase II Step II
Started | 2 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase I
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 66.5 [56 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of FGFR Inhibitor AZD4547
Description: A total of 3 dose levels of AZD4547 were planned: 40mg (level 1), 60mg (level 2), and 80mg (level 3) in combination with a standard dose of docetaxel (75mg/m^2). The starting dose level of AZD4547 was 40 mg. This portion of the study used a standard 3+3 design with patients enrolled in cohorts of 3. The plan was to recommend the maximum tolerated dose (MTD) as the dose level to be used in the phase II portion of the study. MTD is defined as the highest dose level at which less than or equal to 1 of 6 subjects experience dose limiting toxicity (DLT).
Time Frame: Assessed during cycle 1 (21 days)
Measure: Number; unit: mg
Arm/Group | Phase I
Number analyzed (Participants) | 2
mg | NA — As the first two patients experienced DLTs at the lowest dose level of the study, the MTD could not be identified and the study was then closed after having met the predefined criteria for closure per study design.

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment.
Description: Submission of late adverse events is required at follow-up visits up to 3 years.
Arm/Group | Phase I
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I (N=2)
Anemia (Blood and lymphatic system disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Multi-organ failure (General disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Mucosal infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Somnolence (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I (N=2)
Anemia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 2
Edema limbs (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Mucosal infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less